CLINICAL TRIAL: NCT04300660
Title: POPARTS Study- Post-Operative Pain After Recovery in Thoracic Surgery: Evaluation of the Persistence of Painful Symptoms and the Incidence of Neuropathic Pain After Resective Lung Surgery
Brief Title: Post-Operative Pain After Recovery in Thoracic Surgery
Acronym: POPARTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Marzia Umari, Principal Investigator, University of Trieste
Other Study IDs: N. ASUI TS 8/2017
Record Dates: First submitted 2020-03-01; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Neuropathic Pain; Post Operative Pain; Thoracic Surgery
Keywords: thoracic surgery; analgesia; chest wall analgesia; Post-Thoracotomic Pain Syndrome; VATS
MeSH Terms: conditions — Neuralgia; Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: neuropathic pain after thoracic surgery — analysis of perioperative factors implicated in the onset of postoperative pain after chest surgery and the incidence of neuropathic pain

SUMMARY:
Persistent pain after surgery has significant physical and mental consequences for the patient, as well as a significant economic impact on health systems. Neuropathic pain is caused by direct or indirect damage to the somatosensitive system. In thoracic surgery, chronic neuropathic pain is represented by Post-Thoracotomic Pain Syndrome (PTPS), defined as recurrent or persistent pain in the thoracotomy scar site that persists for more than 3-6 months. Currently, in literature, the prevalence of PTPS is extremely variable. This prospective observational study aims to assess the incidence of pain in the weeks and months following surgery and to assess whether and how the presence of painful symptoms changes the patient's quality of life.

DETAILED DESCRIPTION:
For each patient enrolled in the study, in the pre-operative phase, comorbidities, any chronic analgesic therapy and quality of life (through a dedicated questionnaire - Euro QoL 5D5L1) will be recorded. Surgical data (type of procedure, lobe affected by resection, type of approach and surgical time) and anesthesiological data (intravenous opioid, locoregional technique (s), non-opioid analgesics administered and other medications) will be collected in the perioperative phase. In the 48 hours following the surgery (in the Recovery Room, at 6h, 12h, 24h, 36h and 48h) the patient's pain data will be recorded (static, dynamic and cough-associated NRS) and those relating to any complications. The total amount of morphine administered to the patient in the first 48 hours will also be recorded. Each patient will be evaluated 7 days, 1, 3 and 6 months after the surgery by telephone interview. In this last phase, the possible presence of pain and its characteristics will be assessed, especially if these meet the criteria of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient's consent to the trial
* Candidate to resective lung surgery (lobectomy, segmentectomy, atypical resection) with minimally invasive approach (mini-thoracotomy with muscle sparing or video-assisted thoracic surgery, VATS)

Exclusion Criteria:

* neurological and / or cognitive deficits
* inability to obtain informed consent
* surgeries that include wall resections (pleural, muscle, rib or nerve)
* pneumonectomy
* Previous thoracic surgery at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted at our surgical center who underwent elective lobectomy, segmentectomy or atypical resection surgery with a mini-thoracotomy approach or VATS.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of persistent post-operative pain after thoracic surgery | the data needed to analyze the incidence and characteristics of pain will be collected at 1 week after surgery
  The incidence of static, dynamic and cough-associated pain is assessed through the numerical rate scale (NRS), by a telephone interview one week and one month after surgery. A questionnaire is submitted to the patient to analyze the characteristics of the pain and its possible impact on the patient's quality of life.
Incidence of persistent post-operative pain after thoracic surgery | the data needed to analyze the incidence and characteristics of pain will be collected at 1 month after surgery
  The incidence of static, dynamic and cough-associated pain is assessed through the numerical rate scale (NRS), by a telephone interview one week and one month after surgery. A questionnaire is submitted to the patient to analyze the characteristics of the pain and its possible impact on the patient's quality of life.
Incidence of Chronic Pain after thoracic surgery | The data needed to analyze the presence of chronic pain will be collected at 3 months after surgery
  The possible presence and incidence of chronic pain is assessed through a telephone interview three and six months after surgery.
Incidence of Chronic Pain after thoracic surgery | The data needed to analyze the presence of chronic pain will be collected at 6 months after surgery
  The possible presence and incidence of chronic pain is assessed through a telephone interview three and six months after surgery.
Presence of pain with typical features of neuropathic pain in the different phases of the postoperative course | The data neede to analyze the presence of neuropathic pain will be collected at a week after the surgery
  During each telephone interview the presence of neuropathic pain is assessed through a dedicated questionnaire (PainDetect Questionnaire) and the impact that this type of pain has on the patient's quality of life.
Presence of pain with typical features of neuropathic pain in the different phases of the postoperative course | The data neede to analyze the presence of neuropathic pain will be collected at a month after the surgery
  During each telephone interview the presence of neuropathic pain is assessed through a dedicated questionnaire (PainDetect Questionnaire) and the impact that this type of pain has on the patient's quality of life.
Presence of pain with typical features of neuropathic pain in the different phases of the postoperative course | The data neede to analyze the presence of neuropathic pain will be collected at 3 months after the surgery
  During each telephone interview the presence of neuropathic pain is assessed through a dedicated questionnaire (PainDetect Questionnaire) and the impact that this type of pain has on the patient's quality of life.
Presence of pain with typical features of neuropathic pain in the different phases of the postoperative course | The data neede to analyze the presence of neuropathic pain will be collected at 6 months after the surgery
  During each telephone interview the presence of neuropathic pain is assessed through a dedicated questionnaire (PainDetect Questionnaire) and the impact that this type of pain has on the patient's quality of life.

SECONDARY OUTCOMES:
Assessment of the incidence of chronic pain based on the different surgical techniques in thoracic surgery | during the intraoperative phase, data relating to the surgical techniques performed are collected
  the aim of this objective is to analyze whether different surgical techniques (more or less invasive) play a role in the onset of chronic pain after thoracic surgery
Assessment of the post-operative quality of life based on the different surgical techniques in thoracic surgery | during the intraoperative phase, data relating to the surgical techniques performed are collected
  the aim of this objective is to analyze whether different surgical techniques (more or less invasive) play a role in the quality of life after thoracic surgery
Evaluation of postoperative pain control based on different anesthesiological techniques and its possible correlation with the development of chronic pain | data relating to this objective are collected in the intraoperative, 24 hours after surgery and subsequent telephone interviews at 1 week, 1, 3 and 6 months after thoracic surgery
  the aim of this objective is to analyze whether different anesthesiological techniques play a role in the onset of chronic or neuropathic pain after thoracic surgery. The techniques of locoregional anesthesia performed and the drugs used both during surgery and in the postoperative phase are analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Lucangelo, MD PhD, Study Director — University of Trieste; Marzia Umari, MD, Principal Investigator — University of Trieste
Locations (1):
- Cattinara Hospital, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Allegri M, Baron R, Hans G, Correa-Illanes G, Mayoral Rojals V, Mick G, Serpell M. A pharmacological treatment algorithm for localized neuropathic pain. Curr Med Res Opin. 2016;32(2):377-84. doi: 10.1185/03007995.2015.1129321. PMID 26641136
- [Background] Elmore B, Nguyen V, Blank R, Yount K, Lau C. Pain Management Following Thoracic Surgery. Thorac Surg Clin. 2015 Nov;25(4):393-409. doi: 10.1016/j.thorsurg.2015.07.005. PMID 26515940
- [Background] Maguire MF, Ravenscroft A, Beggs D, Duffy JP. A questionnaire study investigating the prevalence of the neuropathic component of chronic pain after thoracic surgery. Eur J Cardiothorac Surg. 2006 May;29(5):800-5. doi: 10.1016/j.ejcts.2006.02.002. Epub 2006 Apr 3. PMID 16581259
- [Background] Rizk NP, Ghanie A, Hsu M, Bains MS, Downey RJ, Sarkaria IS, Finley DJ, Adusumilli PS, Huang J, Sima CS, Burkhalter JE, Park BJ, Rusch VW. A prospective trial comparing pain and quality of life measures after anatomic lung resection using thoracoscopy or thoracotomy. Ann Thorac Surg. 2014 Oct;98(4):1160-6. doi: 10.1016/j.athoracsur.2014.05.028. Epub 2014 Jul 31. PMID 25086945
- [Background] Kinney MA, Mantilla CB, Carns PE, Passe MA, Brown MJ, Hooten WM, Curry TB, Long TR, Wass CT, Wilson PR, Weingarten TN, Huntoon MA, Rho RH, Mauck WD, Pulido JN, Allen MS, Cassivi SD, Deschamps C, Nichols FC, Shen KR, Wigle DA, Hoehn SL, Alexander SL, Hanson AC, Schroeder DR. Preoperative gabapentin for acute post-thoracotomy analgesia: a randomized, double-blinded, active placebo-controlled study. Pain Pract. 2012 Mar;12(3):175-83. doi: 10.1111/j.1533-2500.2011.00480.x. Epub 2011 Jun 16. PMID 21676165
- [Background] Gotoda Y, Kambara N, Sakai T, Kishi Y, Kodama K, Koyama T. The morbidity, time course and predictive factors for persistent post-thoracotomy pain. Eur J Pain. 2001;5(1):89-96. doi: 10.1053/eujp.2001.0225. PMID 11394926
- [Background] Khelemsky Y, Noto CJ. Preventing post-thoracotomy pain syndrome. Mt Sinai J Med. 2012 Jan-Feb;79(1):133-9. doi: 10.1002/msj.21286. PMID 22238046
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849